CLINICAL TRIAL: NCT05001386
Title: Evaluation of Anti-cancer Drugs Sensitivity on Fresh Samples From Healthy Patients and Patients With Myeloproliferative or Lymphoproliferative Disorders
Brief Title: In Vitro Drug Sensitivity Testing of Fresh Human Samples
Acronym: ESAAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_0622
Record Dates: First submitted 2021-07-27; First posted 2021-08-11 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Myeloproliferative Disorders; Lymphoproliferative Disorders
Keywords: Hematological malignancies; lymphoid; myeloid; multiple myeloma; anticancer drugs; sensitivity; new treatments
MeSH Terms: conditions — Myeloproliferative Disorders; Lymphoproliferative Disorders; Hematologic Neoplasms; Multiple Myeloma; Hypersensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lymphoproliferative disorders (Experimental): Patients followed in the haematology unit of Hospices Civils de Lyon for lymproliferative disorders as chronic lymphoid leukemia (CLL), non-Hodgkin lymphoma (NHL) or multiple myeloma (MM) .
  Interventions: Biological: Blood collection for the evaluation of the anti-drugs sensitivity
- Control group (Sham Comparator): Patients followed in the medicine of aging unit in the Hospices Civils de Lyon without haematological malignancies, without chemotherapy and without immunosuppressive treatment (≤ 5 years)
  Interventions: Biological: Blood collection for the evaluation of the anti-drugs sensitivity
- Myeloproliferative disorders (Experimental): Patients followed in the haematology unit of Hospices Civils de Lyon for myeloproliferative disorders as acute myeloid leukemia (AML) or chronic myeloid leukemia (CML).
  Interventions: Biological: Blood collection for the evaluation of the anti-drugs sensitivity

INTERVENTIONS:
Biological: Blood collection for the evaluation of the anti-drugs sensitivity — The M.D investigators and the medical team identify the patients ( index cases and healthy volunteers) in a medical appointment. They inform them, collect the non-opposition right and the blood samples: 5 mL heparin tube and 5 mL dry tube for each person , one time.

SUMMARY:
Hematological malignancies gather several various pathologies included myeloproliferative disorders (as acute myeloid leukemia (AML) or chronic myeloid leukemia (CML)) and lymphoproliferative disorders (as chronic lymphoid leukemia (CLL), non-Hodgkin lymphoma (NHL) and multiple myeloma (MM)) .

Over the last decade, the treatments have evolved significantly but the overall survival remains limited, especially for the AML and MM patients. There's an ongoing imperative to continue in-vitro and in-vivo studies to better evaluate the anti-cancer drugs sensitivity and therefore improving the response to treatments and open new fields of application. The healthy control group will be contributing to produce some pertinent and significant data for the results of the index cases group.

The investigators aim to analyze 10 differents drugs, common use in chemotherapy or immunotherapy and evaluate by 2 ways the sensitivity: first, Flow cytometry (cells apoptosis by Annexine V and propidium iodide) on fresh samples and in a second time, monitoring of the blasts in the mouse's blood after injection.

ELIGIBILITY:
Inclusion Criteria:

* Index cases: patients with myeloproliferative or lymphoproliferative disorders.
* Controls: patients without hematological disease, without chemotherapy ((≤ 5 years.) and without immunosuppressive treatment at the study time.
* Age ≥ 18 y.o for all the patients

Exclusion Criteria:

* Age < 18 y.o
* Pregnant or breastfeeding woman
* Patients deprived of their liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the sensitivity of 10 anti-cancer drugs | Through study completion, an average of 3 years
  Sensitivity determined by in-vitro
  * Tumor cells mortality by Flow cytometry
  * Monitoring of the blasts in the mouse's blood after injection
Evaluation of the sensitivity of 10 anti-cancer drugs | Through study completion, an average of 3 years
  Sensitivity determined by in-vivo fresh samples:

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Lyon Sud -Service d'Hématologie, Pierre-Bénite
  - Centre Hospitalier Lyon Sud -Service de médecine du vieillissement, Pierre-Bénite